CLINICAL TRIAL: NCT02447744
Title: Neural Changes Associated With a Mindfulness-based Intervention for Young Adults With Childhood Maltreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Sara W Lazar, Associate Research Scientist, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000295
Record Dates: First submitted 2014-12-02; First posted 2015-05-19 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Depression; Anxiety; PTSD; Trauma, Psychological
Keywords: depression; anxiety; childhood trauma; mindfulness
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Psychological Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness group (Experimental): This arm receives an 8-week mindfulness based behavioral intervention program.
  Interventions: Behavioral: Mindfulness based intervention
- Waitlist control group (Other): This arm waits while the mindfulness group receives their intervention, and then receives the mindfulness based intervention after their waiting period.
  Interventions: Behavioral: Mindfulness based intervention

INTERVENTIONS:
Behavioral: Mindfulness based intervention — The intervention is an 8-week structured mindfulness based behavioral intervention program that teaches mindfulness meditation, mindful yoga and psychological knowledge about stress.

SUMMARY:
Childhood trauma is remarkably prevalent, and it has long lasting impact on mental health and neural development. This trial aims to see whether the 8-week mindfulness based intervention can reduce stress related psychological symptoms for young adults with childhood maltreatment, and whether it can promote neural plasticity.

DETAILED DESCRIPTION:
This study recruits young adults with childhood adversity; enrolled subjects either receive an 8-week mindfulness based intervention, or wait for 8 weeks before receiving the intervention. MRI and a battery of self report questionnaires will be administered before and after the intervention; subjects on the waiting list will undergo the same research procedures at the same time as subjects in the intervention group. Primary hypotheses include improved hippocampal plasticity, increased mindfulness and reduced stress and related psychological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Experience of childhood maltreatment
* With current age between 19 to 35 years old
* With current symptoms of depression or anxiety or PTSD or significant general stress.

Exclusion Criteria:

* History of psychiatric disorders with psychotic features
* Suicidal attempts during the past six months
* Neurological disorders
* And common MRI exclusion criteria
* Prior history with the mindfulness based stress reduction program or other systematic meditation programs.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-07-21 (Actual); Study Completion 2016-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lazar, PhD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Joss D, Khan A, Lazar SW, Teicher MH. Effects of a Mindfulness-Based Intervention on Self-Compassion and Psychological Health Among Young Adults With a History of Childhood Maltreatment. Front Psychol. 2019 Oct 23;10:2373. doi: 10.3389/fpsyg.2019.02373. eCollection 2019. PMID 31749731

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness Group | Waitlist Control Group
Started | 21 (6 subjects are enrolled in the mindfulness program after serving on the waiting list control group) | 22
Completed | 15 | 21
Not Completed | 6 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Data not collected b/c logistic reasons | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Group | Waitlist Control Group | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Full Range); unit: years] | 26.667 [22 to 34] | 25.273 [22 to 29] | 25.953 [22 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 12 | 16 | 28
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Changes in Subjects' Perceived Stress Level
Description: Changes in the Perceived Stress Scale scores (post- intervention scores minus pre- intervention scores). Relevant time points used in the calculation include baseline scores at enrollment, and post-intervention/waiting period scores after 2 months of intervention or waiting period. Calculations of the change entail post-intervention/waiting period scores minus baseline scores for each individual subject.
  The Perceived Stress Scale is a 10 item scale (each responded with Likert scale 0-4), the scale score is the sum of all items, thus the full range of PSS scores is 0-40, with higher scores means worse stress. A reduction in PSS scores (i.e., the change scores being negative) indicates subjects have improved after the intervention by becoming less stressed.
Time Frame: After the 8-week intervention program compared to baseline measurement, or the same time as the intervention group for subjects on the waiting list.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Group | Waitlist Control Group
Number analyzed (Participants) | 19 | 17
score on a scale | -5.526 (1.566) | 1.000 (1.437)

2. Secondary Outcome: Changes of Mindfulness
Description: Changes in the mindfulness level as measured by the Mindful Attention Awareness Scale (post-intervention scores minus pre-intervention scores).
  Relevant time points used in the calculation include baseline scores at enrollment, and post-intervention/waiting period scores after 2 months of intervention or waiting period. Calculations of the change entail post-intervention/waiting period scores minus baseline scores for each individual subject.
  The MAAS is a 15-item scale each responded with Likert scale 1-6; the MAAS score calculated as the mean of all items, thus the full range of the score is 1-6, with higher scores meaning more mindful. An increase in MAAS score (i.e., a positive score change )means the subject has improved after the intervention by becoming more mindful.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Group | Waitlist Control Group
Number analyzed (Participants) | 18 | 15
score on a scale | 0.337 (0.149) | 0.049 (0.126)

3. Post Hoc Outcome: Percent Changes of Right Hippocampal Grey Matter Density
Description: Gray matter density of the right hippocampus is calculated from anatomical MRI data with the SPM software. Percent changes of gray matter density is calculated for each subject. Relevant time points used in the calculation include baseline values at enrollment, and post-intervention/waiting period values after 2 months of intervention or waiting period. Calculations of the change entail post-intervention/waiting period values minus baseline values, then divided by the baseline values to obtain the percent change measure.
Time Frame: 2 months
Population: Subjects who completed both baseline and post-intervention/waiting period were entered into analyses. 6 Subjects from the waiting list control group completed a third MRI after completing the mindfulness intervention.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Mindfulness Group | Waitlist Control Group
Number analyzed (Participants) | 21 | 21
Percent change | 0.8137 (0.3143) | -0.9229 (0.2014)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between the period of time when subjects are enrolled in the study and when subjects complete the post-intervention research procedures, or till subjects voluntarily drop out of the study before the completion of intervention and research procedures. The time frame is up to 2 years.
Arm/Group | Mindfulness Group | Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No